CLINICAL TRIAL: NCT00579813
Title: Mechanisms Underlying Metabolic Syndrome in Obesity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Philip Kern (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Philip Kern, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 32677; R01DK071277 (NIH)
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Results first posted 2011-07-12 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-05

CONDITIONS: Metabolic Syndrome; Insulin Resistance; Prediabetes
Keywords: obesity; inflammation; diabetes
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Prediabetic State; Obesity; Inflammation; Diabetes Mellitus | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 (No Intervention): Baseline studies (OGTT, DXA, RMR, FSIGT, and biopsies) on normal control subjects. Oral glucose tolerance tests, body composition assessment, resting metabolic rate, insulin sensitivity measurement with the frequently sampled method and Minimal Model. These studies will establish baseline data in lean subjects on adipose tissue gene expression, insulin sensitivity, glucose tolerance, metabolic rate and body composition. There is no intervention.
- 2 (Active Comparator): Baseline studies (OGTT, DXA, RMR, FSIGT, biopsies), then 10 weeks treatment on Pioglitazone. Baseline tests are repeated at the end of medication treatment. All of the studies described in arm 1 are repeated after treatment. The subjects in this group have impaired glucose tolerance. After the measurement of adipose tissue gene expression, insulin sensitivity, glucose tolerance, metabolic rate and body composition, subjects are treated with pioglitazone, working up to 45 mg/day, for 10 weeks. After this time, adipose tissue gene expression, insulin sensitivity, glucose tolerance, metabolic rate and body composition are repeated.
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone 30mg for 2 weeks, then Pioglitazone 45mg for 8 weeks.
  Other Names: Actos
  Arms: 2

SUMMARY:
The purpose of this study is to better understand the link between obesity and diabetes or pre-diabetes.

DETAILED DESCRIPTION:
Obesity is the most common and powerful force for creating insulin resistance and metabolic syndrome, however, the molecular basis of this association is not well understood. In this proposal, three independently funded researchers-Philip Kern, MD a clinical investigator, and Charlotte Peterson, PhD and Robert McGehee, PhD, with significant experience in muscle and adipocyte biology, respectively-will formalize a collaborative effort as a natural extension of previous work and shared interests in the fields of obesity, insulin resistance, and tissue lipid accumulation. Our overall hypothesis is that insulin resistance in humans stems largely from ectopic accumulation of intramyocellular lipid (IMCL) during the development of obesity. Further, we hypothesize that excess IMCL accumulation is dependent on secretory proteins derived from a complex interplay between adipocytes and macrophages in adipose tissue. To test these hypotheses, we will examine the interactions among adipocytes, macrophages, and muscle cells isolated and cultured from subjects that are obese with insulin resistance and impaired glucose tolerance (IGT), and from some with Type 2 Diabetes. This study population has elevated IMCL and is at high risk for obesity complications, but avoids the pathophysiologic complications of glucotoxicity. These subjects will be compared to obese subjects with normal glucose tolerance (NGT).

Aim 1 will explore mechanisms that contribute to IMCL and elucidate its role in the development of IGT. Cultured muscle cells will be used to determine whether obese subjects with IGT versus NGT demonstrate intrinsic differences in muscle gene expression and metabolic activity under differing extracellular fatty acid concentrations. Lipid accumulation and oxidation, and insulin-mediated glycogen synthesis and signaling will be assessed.

Aim 2 will determine if the IMCL accumulation is dependent on adipose tissue secretory proteins. We will use co-cultures of adipocytes, myoblasts, and adipose stromal vascular cells to examine IMCL and the development of insulin resistance.

Aim 3 will determine whether the stromal fraction from IGT subjects promotes IMCL more effectively than that from NGT subjects in co-cultures with muscle cells. We will compare the stromal vascular fractions with regard to monocyte/macrophage accumulation and cytokine expression.

Aim 4 will determine if improved glucose tolerance in response to a 10-week treatment with pioglitazone results in decreased IMCL and identify cellular mechanisms involved. Co-culture studies will also be used with muscle and stromal cells, before and after pioglitazone treatment. These experiments will provide mechanistic insight into the link between obesity and muscle function leading to metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* BMI 28+
* diabetes, impaired glucose tolerance or normal glucose tolerance

Exclusion Criteria:

* AST >2x normal
* congestive heart failure
* history of coronary artery disease
* chronic renal insufficiency (creatinine > 1.4mg/dl)
* use of gemfibrozil, ACE inhibitors, and angiotensin receptor II blockers, or anticoagulants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2005-04; Primary Completion 2009-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Kern, MD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of Kentucky, Lexington, Kentucky

IPD SHARING:
Plan to Share IPD: Yes
Data from this study has been published. Individual (deidentified) data will be shared with other investigators upon request to Dr Kern.

RESULTS

PARTICIPANT FLOW:
Groups:
- Lean Subjects: Arm 1 was normal subjects on which baseline studies were performed to determine insulin sensitivity, intramyocellular lipid and resting metabolic rate.
- Obese Subjects: Baseline studies (Oral glucose tolerance test, Dual energy x-ray absorbiometry, Resting metabolic rate, Frequently sampled intravenous glucose tolerance test, biopsies), then 10 weeks treatment on Pioglitazone. Baseline tests are repeated at the end of medication treatment.
Period: Overall Study
Arm/Group | Lean Subjects | Obese Subjects
Started | 60 | 10
Completed | 60 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lean Subjects | Obese Subjects | Total
Number analyzed (Participants) | 60 | 10 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 10 | 70
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (6) | 57 (2) | 55 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 7 | 52
  Male | 15 | 3 | 18
Region of Enrollment [Number; unit: participants]
  United States | 60 | 10 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulin Sensitivity Using FSIGT
Description: The frequently sampled intravenous glucose tolerance test (FSIGT) involves the injection of IV glucose and the frequent measurement of glucose and insulin.
Time Frame: Baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: FSIGT units (x10^-4/min/uU/ml)
Groups:
- Obese Subjects, Baseline: Baseline studies, obese
- After Pioiglitazone: 10 weeks of treatment
- Lean Subjects, Baseline: lean subjects, baseline
Arm/Group | Obese Subjects, Baseline | After Pioiglitazone | Lean Subjects, Baseline
Number analyzed (Participants) | 10 | 10 | 60
FSIGT units (x10^-4/min/uU/ml) | 1.7 (0.53) | 2.4 (1.01) | 7.02 (3.7)

2. Primary Outcome: Effects of Pioglitazone on Changes in BMI
Description: Body Mass Index (BMI) is measured at baseline, in lean and obese subjects, and after pioglitazone in obese subjects
Time Frame: Baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Obese Subjects, Baseline | After Pioiglitazone | Lean Subjects, Baseline
Number analyzed (Participants) | 10 | 10 | 60
kg/m2 | 32.4 (3.89) | 33.4 (4.36) | 22.6 (1.9)

3. Primary Outcome: Changes in Muscle Lipid After Pioglitazone
Description: Muscle lipid following biopsy using oil red-O staining.
Time Frame: At baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: arbitrary units of oil red O staining
Arm/Group | Obese Subjects, Baseline | After Pioiglitazone | Lean Subjects, Baseline
Number analyzed (Participants) | 10 | 10 | 60
arbitrary units of oil red O staining | 7.0 (5.9) | 4.6 (5.9) | 2.7 (0.84)

4. Primary Outcome: Changes in Fat Inflammation Following Pioglitazone
Description: macrophages in fat at baseline, in lean and obese participants, and obese after pioglitazone (in obese)
Time Frame: Baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: macrophages per mm2 by CD68 staining
Arm/Group | Obese Subjects, Baseline | After Pioiglitazone | Lean Subjects, Baseline
Number analyzed (Participants) | 10 | 10 | 60
macrophages per mm2 by CD68 staining | 27 (6.3) | 19 (9.5) | 17 (6.2)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Lean Subjects | Obese Subjects
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/10
Other Adverse Events (participants affected / at risk) | 0/60 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No